CLINICAL TRIAL: NCT00048256
Title: Exploring the Relationship Between Personality and Coping Styles in Bone Marrow Transplant Candidates
Brief Title: Relationship Between Personality and Coping Styles in Bone Marrow Transplant Candidates
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030028; 03-CC-0028
Record Dates: First submitted 2002-10-28; First posted 2002-10-29 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-09

CONDITIONS: Adaptation, Psychological; Bone Marrow Transplantation
Keywords: Cancer; Personality Assessment; Coping Styles; Psychological Distress; Bone Marrow Transplants; Bone Marrow Transplant
MeSH Terms: conditions — Neoplasms

SUMMARY:
This study will look at how people cope with an upcoming bone marrow transplant and how personality characteristics influence coping styles in stressful medical situations. Personality traits, such as extraversion, optimism and self-esteem have been related to active, problem-focused coping styles, whereas neuroticism has been related to increased psychological distress and denial as a way of coping. Coping styles, in turn, have been related to disease outcome. For example, a fighting spirit and avoidance have been correlated with longer survival, whereas fatalism, anxious preoccupation and feelings of helplessness and hopelessness were related to a poor disease outcome. A better understanding of the relationship between coping styles and personality may help improve supportive care for people undergoing bone marrow transplants. This study will:

* Explore the relationship between personality traits, coping styles and psychological stress in patients awaiting bone marrow transplantation
* Identify what coping styles people use to prepare for bone marrow transplantation
* Identify what personality traits are related to particular coping styles in patients awaiting bone marrow transplantation
* Identify the relationship between personality factors and level of psychological distress in patients awaiting bone marrow transplantation

Cancer patients 18 years of age and older who are scheduled for bone marrow transplant are eligible for this study.

Participants will fill out pencil-and-paper questionnaires providing demographic information (such as age, gender, marital status, ethnicity, and so forth) and answering questions about their opinions and preferences. The information will be used to assess the participants' personality characteristics, coping styles, and psychological distress. The questionnaires take about 45 to 50 minutes to complete.

DETAILED DESCRIPTION:
Over the last decade, more and more focus has been placed upon the psychological adjustment of patients who have undergone bone marrow transplants (BMT). There have been studies that focused on the coping styles and levels of psychological distress in patients immediately after transplantation. Studies have been done based on a specific point during the process or at multiple points throughout the course of the procedure and still other studies have focused on assessment points several months post transplant. However, very little attention has been focused on patients' psychological functioning prior to transplantation. The purpose of the present study is to examine the relationship between personality traits and coping styles among patients awaiting BMT.

ELIGIBILITY:
INCLUSION CRITERIA

All patients with diagnosis of cancer and awaiting BMT.

Criteria for participation in the study include a diagnosis of cancer and being actively screened for a CC approved PBSC transplant protocol. The participants will not have undergone the transplant at the time of the evaluation. Participants will be ages 18 and older.

EXCLUSION CRITERIA

No patients who meet the eligibility criteria will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57
Dates: Start 2002-10; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center (CC), Bethesda, Maryland, United States